CLINICAL TRIAL: NCT00678184
Title: The Effect of Acute HMG-CoA-Reductase Inhibition (Atorvastatin) on Renal Sodium Excretion, Renal Hemodynamics, Tubular Function and Vasoactive Hormones in Healthy Subjects During Normal and High Sodium Intake
Brief Title: The Effect of Atorvastatin on Renal Function in Healthy Subjects During Normal and High Sodium Intake
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MED.RES.HOS.2006.03.LP
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Last update posted 2008-05-15 (Estimated); Status verified 2008-05

CONDITIONS: Healthy Subjects
Keywords: Atorvastatin; healthy; sodium excretion; hemodynamics; tubular function
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Atorvastatin — 80 mg atorvastatin on two following days each

SUMMARY:
We wanted to test the hypothesis that acute treatment with atorvastatin changes renal sodium handling, renal hemodynamics, tubular function and vasoactive hormones in healthy humans during normal and high sodium intake.

DETAILED DESCRIPTION:
We wanted to test the hypothesis that acute treatment with atorvastatin changes renal sodium handling, renal hemodynamics, tubular function and vasoactive hormones in healthy humans during normal and high sodium intake.

We wanted to analyze if changes in renal hemodynamics, tubular function, hormones, blood pressure and HR under acute treatment with atorvastatin depends on sodium intake.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-50 yr
2. BMI<30
3. Females had to use oral contraceptive treatment or IUD.

Exclusion Criteria:

1. Clinical signs or history of disease of the heart, lungs, kidneys, liver, brain or endocrine organs
2. Abnormal laboratory blood tests (hemoglobin, sodium, potassium, albumin, creatinine, blood glucose, bilirubin, alanin amino transferase, alkalic phosphatase)
3. Albuminuria or glucosuria
4. cancer
5. arterial hypertension
6. alcohol abuse
7. medical treatment, except contraceptives
8. pregnancy or breast feeding
9. blood donation one month before the study.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2007-01; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Glomerular filtration rate, clearance of sodium and lithium, fractional excretion of sodium and lithium, U-AQP-2, total sodium excretion, free water clearance | 6 months

SECONDARY OUTCOMES:
AVP, Ang-II, Aldosterone, ANP, BNP, PRC, BP and HR. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Erling B. Pedersen, Professor, Principal Investigator — Dept. of medical reaserch, Holstebro Hospital, Denmark
Locations (2):
- Denmark (2):
  - Department of Medical Research, Holstebro Hospital, Holstebro
  - Medical Research, Holstebro